CLINICAL TRIAL: NCT03537482
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Property of Orally Administered APG-2575 in Patients With Hematologic Malignancies
Brief Title: APG-2575 Study of Safety, Tolerability ,PK/PD in Patients With Hematologic Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG2575-001
Record Dates: First submitted 2018-03-27; First posted 2018-05-25 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Lisaftoclax

STUDY DESIGN:
Intervention Model Description: dose escalation and dose expansion after MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single-agent, open-label, Phase I study of APG-2575 (Experimental): The study consists of the dose escalation stage and the dose expansion stage
  Interventions: Drug: APG-2575

INTERVENTIONS:
Drug: APG-2575 — APG-2575 will be administered as an oral tablet

SUMMARY:
This is a multi-center, single-agent, open-label, Phase I study of APG-2575. The study consists of the dose escalation stage and the dose expansion stage.

DETAILED DESCRIPTION:
APG-2575 will be administered orally, once daily for consecutive 4 weeks as one cycles. Initially, the start dose is 20mg. Single patient cohorts will be evaluated, the dose of APG-2575 will be increased in subsequent cohorts, to 50 mg, 100 mg, 200 mg, 400 mg, 600mg and 800mg accordingly. If there is any one of the following event is observed, a DLT, two drug related Grade 2 toxicities or one drug related ≥ Grade 3 toxicity, or laboratory or clinical TLS, or suspected hypersensitivity reaction occur in Cycle 1, or dose level of 400 mg is reached, the dose escalation will convert to the standard 3+3 design, If ≥ 2/6 patients develop DLT at any dose level dose escalation will cease and the dose level immediately below will be expanded to 6 patients. If ≤ 1/6 patients develop a DLT at the highest dose reached this will be declared the MTD. After the MTD is defined, a maximum of 20 patients will be treated at that dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Histologically confirmed diagnosis of either one of the B-cell hematologic malignancies including multiple myeloma, chronic lymphocytic leukemia, lymphoplasmacytic lymphoma, and non-Hodgkin's lymphoma such as mantle cell lymphoma, diffuse large B cell lymphoma, Waldenstrom macroglobulinemia (WM) and acute myeloid leukemia
3. Patient must have relapsed or refractory to, intolerant to, or are considered ineligible for therapies known to provide clinical benefit. In addition,

   a. AML Patients will be eligible if they have failed standard induction regimen, are not considered candidate for further chemotherapy or stem cell transplantation or have primary refractory AML.
4. Life expectancy ≥ 3 months.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 -1 in dose escalation ; 0-2 in dose expansion.
6. QTc interval ≤450ms in males, and ≤470ms in females.
7. Adequate bone marrow function independent of growth factor:
8. Absolute neutrophil count (ANC) ≥1.0 X 109/L.
9. Hemoglobin ≥ 8.0 g/dL.
10. Platelets count ≥ 30 X 109/L (entry platelet count must be independent of transfusion within 7 days of first dose).
11. Adequate renal and liver function as indicated by:

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Prior history of allogeneic cell transplant.
2. Subjects have been diagnosed with Burkitt's lymphoma, Burkitt-like lymphoma, or lymphoblastic lymphoma/leukemia.
3. Received chemotherapy within 14 days (42 days for nitrosoureas or mitomycin C) prior to entering the study.
4. Received biologic (< 28 days), small molecule targeted therapies (< 5 half-life) or other anti-cancer therapy within 21 days of study entry.
5. Radiation within 14 days of study entry, thoracic radiation within 28 days of study entry.
6. Has gastrointestinal conditions that could affect the absorption of APG-2575 in the opinion of the Investigator.
7. Has known active central nervous system (CNS) involvement.
8. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 1 except alopecia or neuropathy.
9. Concurrent treatment with an investigational agent, 14 days for small molecular agents and/or 28 days for biologics treatment prior to the first dose of therapy.
10. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients with active wound healing, patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
11. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
12. Active rheumatoid arthritis (RA), active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation.
13. Active infection requiring systemic antibiotic/ antifungal medication, known clinically active hepatitis B or C infection, or on antiretroviral therapy for HIV disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Patients with APG-2575 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 4.0

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  Maximum plasma concentration (Cmax) will be assessed in the patients treated with APG-2575
Area under the plasma concentration versus time curve (AUC) | 28 days
  Area under the plasma concentration versus time curve (AUC) of APG-2575 will be assessed in the patients treated with APG-2575
Anti-tumor effects of APG-2575 | up to 2 years
  Response will be evaluated every 2 cycles (8 weeks), by the investigator based on disease specific criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (5):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Duke Unviersity, Durham, North Carolina
  - MDACC, Houston, Texas
- Australia (2):
  - St. Vincent Hospital, Fitzroy, Victoria
  - Epworth Healthcare, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: No